CLINICAL TRIAL: NCT01307150
Title: Evaluation of the Efficacy of Dead Sea Climatotherapy on Atopic Dermatitis Patients.
Brief Title: Climatotherapy At The Dead Sea For Atopic Dermatitis
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: Hasassah Medical Organization IRB, Israel Ministry of Health
Other Study IDs: SK09409-HMO-CTIL
Record Dates: First submitted 2009-07-06; First posted 2011-03-02 (Estimated); Last update posted 2011-03-02 (Estimated); Status verified 2009-07

CONDITIONS: Atopic Dermatitis
Keywords: Atopic Dermatitis; Dead Sea; Climatotherapy; SCORAD
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Before and after treatment: SCORAD of each patient before and after treatment.

SUMMARY:
The purpose of this study is to evaluate the improvement in severity of Atopic Dermatitis and quality of life after 4 weeks of treatment in the Dead Sea.

DETAILED DESCRIPTION:
28 days treatment period, sun exposure and possibly Dead Sea baths after an exact given plan, discontinuation of all local Cortisone preparations, unlimited use of maintenance drags, doctor visit twice a week, continuous checks by the nurse.

Determination of the SCORAD index by the same doctor on arrival and departure. Before and after the treatment, the patient will answer written questionnaires regarding quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Minimum age of 18 years old

Exclusion Criteria:

* Skin type - I
* Psoriasis patient in addition to Atopic Dermatitis
* Pregnancy
* Past malignancy
* Less then 2 weeks of treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Atopic Dermatitis patient.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2009-06; Primary Completion 2009-11 (Estimated); Study Completion 2009-12 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Arie Ingber, MD., Study Chair — Hadassa Medical Organization IRB
Locations (1):
- DMZ Clinic, Jerusalem, Israel

REFERENCES:
- [Result] Harari M, Shani J, Seidl V, Hristakieva E. Climatotherapy of atopic dermatitis at the Dead Sea: demographic evaluation and cost-effectiveness. Int J Dermatol. 2000 Jan;39(1):59-69. doi: 10.1046/j.1365-4362.2000.00840.x. PMID 10651969